CLINICAL TRIAL: NCT04504435
Title: A Randomized, Double-blind, Placebo-controlled, First Time in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single (in Both Fed and Fasted States) Doses of GSK3494245 in Healthy Participants
Brief Title: Safety, Tolerability and Pharmacokinetics (PK) Investigation of GSK3494245 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 208441; 2019-004492-39 (EudraCT Number)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Leishmaniasis
Keywords: GSK3494245; Leishmaniasis; Single Ascending Dose; First Time in Human; Pharmacokinetics
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Intervention Model Description: The study will consist of 3 cohorts (Cohorts 1, 2 and 3), conducted in sequential order. Cohorts 1 and 2 will consist of a single dose, ascending, crossover design. Cohorts 1-2 will comprise of a 4-way crossover which includes 4 dosing regimens under fasted conditions. Cohort 3 will comprise of a 2-way crossover which includes 1 dosing regimen under fasted then fed condition and 1 regimen under fed then fasted condition in a 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study with respect to allocation of GSK3494245 or placebo to participants. The food effect part of the study will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Participants in Cohort 1 (Experimental): Participants will receive a maximum of 3 ascending dose levels of GSK3494245 starting with 20 milligram (mg) and 1 placebo dose orally on Day 1 of each treatment period under fasted conditions. There will be a washout period of at least 48 hours or 5-half-lives (whichever is longer) between each dose for an individual participant.
  Interventions: Drug: GSK3494245; Drug: Placebo
- Participants in Cohort 2 (Experimental): Participants will receive a maximum of 3 ascending dose levels of GSK3494245 starting with dose level (DL) 5 and 1 placebo dose orally on Day 1 of each treatment period under fasted conditions. There will be a washout period of at least 48 hours or 5-half-lives (whichever is longer) between each dose for an individual participant.
  Interventions: Drug: GSK3494245; Drug: Placebo
- Cohort 3: Participants receiving GSK3494245 (fasted then fed) (Experimental): Participants will receive the selected dose level (DLX) of GSK3494245 in the fasted state on Day 1 in Period 1 followed by a single dose of GSK3494245 in the fed state in Period 2. There will be a washout period of at least 48 hours or 5-half-lives (whichever is longer) between each dose for an individual participant.
  Interventions: Drug: GSK3494245
- Cohort 3: Participants receiving GSK3494245 (fed then fasted) (Experimental): Participants will receive the DLX of GSK3494245 in the fed state on Day 1 in Period 1 followed by a single dose of GSK3494245 in the fasted state in Period 2. There will be a washout period of at least 48 hours or 5-half-lives (whichever is longer) between each dose for an individual participant.
  Interventions: Drug: GSK3494245

INTERVENTIONS:
Drug: GSK3494245 — Capsule of 10-250 mg dose strength will be provided in labelled High Density Polyethylene (HDPE) bottles.
Drug: Placebo — Matching placebo capsules will be provided
  Arms: Participants in Cohort 1; Participants in Cohort 2

SUMMARY:
This is a Phase 1, double-blind, randomized, placebo-controlled, first time in human (FTIH) study to assess the safety, tolerability and PK of a single dose of GSK3494245. The study will consist of 3 cohorts, conducted in a sequential manner. Cohorts 1 and 2 will consist of a single ascending dose (SAD), crossover design where each participant will receive a maximum of 3 ascending oral doses of GSK3494245 and 1 placebo dose under fasted conditions. At each dose level, GSK3494245 and placebo will be administered in a 3:1 ratio, within each period, according to the randomization schedule in a blinded manner. Cohort 3 will comprise of a 2-way crossover which includes 1 dosing regimen under fasted then fed conditions and 1 regimen under fed then fasted conditions in a 1:1 ratio. The fed conditions will investigate the effect of safety, tolerability and PK of a single dose of GSK3494245 following food administration.

ELIGIBILITY:
Inclusion Criteria

* Participant must be 18 to <=50 years of age, at the time of signing the informed consent.
* Participant must be healthy as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the normal reference range for the population being studied may be included only if the Investigator in consultation with the Medical Monitor (if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 Kilograms (kg) and body mass index (BMI) within the range 18.5-28 Kilograms per meter square (kg/m^2) (inclusive).
* Male participants only. A male participant with a female partner of reproductive potential must agree to use contraception during the intervention period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed consent form (ICF) and protocol.

Exclusion Criteria

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal blood pressure, as determined by the investigator.
* Previous history of leishmaniasis.
* Alanine aminotransferase (ALT) greater than 1.5 times upper limit of normal (ULN).
* Total bilirubin greater than 1.5 times ULN (isolated bilirubin greater than 1.5 times ULN is acceptable if total bilirubin is fractionated and direct bilirubin less than 35 percent [%]).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or history of clinically significant gastritis or gastroduodenal ulcers or regular use of non-steroidal anti-inflammatory drugs (NSAID).
* Consumption of greater than 14 units/week alcohol (male volunteers).
* Current or history of change in taste or smell without any plausible clinical explanation based on investigator's clinical judgement.
* QTc greater than 450 milliseconds (msec) based on average of triplicate ECGs.
* Waveform abnormalities including premature ventricular contraction (PVC) triplets and more than 500 single PVCs in 24 hours, or any other abnormalities at the discretion of investigator.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Past or intended use of over-the-counter or prescription medication, including herbal medications, NSAIDs, proton pump inhibitors (PPIs) or anti-histamine 2 receptor (H2) antagonists within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longest) prior to dosing. Other concomitant medication may be considered on a case by case basis by the investigator in consultation with the medical monitor. Paracetamol is permitted (capped to <=2 grams/day).
* Participation in the study that would result in loss of blood or blood products in excess of 500 milliliter (mL) within a 56-day period.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study intervention or any other type of medical research.
* Current enrollment or past participation in this clinical study.
* Participants with renal function defined as Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) with an age appropriate Glomerular filtration rate (GFR) <90 (milliliter per minute per 1.73 meter square [mL/min/1.73m^2]).
* Screening urine albumin:creatinine ratio >30 milligram per gram (mg/g) (>3 milligram per millimole [mg/mmol])
* Presence of hepatitis B surface antigen (HBsAg) test result at screening.
* Positive hepatitis C antibody test result at screening.
* Positive hepatitis C Ribonucleic acid (RNA) test result at screening.
* Positive human immunodeficiency virus (HIV) antibody test.
* Presence of clinically significant hematuria and/or proteinuria.
* Carbon monoxide levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 3 months prior to screening.
* Positive pre-study drug/alcohol screen.
* Regular use of known drugs of abuse.
* Food Effect Cohort 3 only: Participant must have no dietary restrictions (e.g., lactose intolerance) or inability to eat gelatin or an adapted standard meal (includes 35-40% fat content).
* Food Effect Cohort 3 only: History of gall bladder surgery or gall bladder removal, or history of an acute disease state (e.g. cholelithiasis) within 14 days prior to receiving the study treatment.
* Participants must not have travelled to an area (as determined by the investigator) with a high prevalence of leishmanial/parasitic infections in the 6 months before screening or intend to do so in the 3 months after the final dose of study treatment.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates participation in the study.
* A positive laboratory confirmation of corona virus disease 2019 (COVID-19) infection, or high clinical index of suspicion for COVID-19.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A male participant with a female partner of reproductive potential must agree to use contraception during the intervention period and for at least 90 days after the last dose of study treatment and refrain from donating sperm during this period.
Enrollment: 59 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | Up to 14 days post last dose in each treatment period
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAE is defined as any untoward medical occurrence that, at any dose: results in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Number of participants with treatment emergent AEs and SAEs | Up to 14 days post last dose in each treatment period
  Treatment emergent AE and SAE are any untoward medical occurrences in a clinical study participant, having causal relation with the use of a study intervention.
Number of participants with clinically significant abnormal findings in hematology parameters | Up to 14 days post last dose in each treatment period
  Blood samples will be collected for the assessment of hematology parameters.
Number of participants with clinically significant abnormal findings in clinical chemistry parameters | Up to 14 days post last dose in each treatment period
  Blood samples will be collected for the assessment of chemistry parameters
Number of participants with urinalysis findings | Up to 14 days post last dose in each treatment period
  Urine samples will be collected for the assessment of urinalysis parameters.
Number of participants with clinically significant abnormal findings in vital signs | Up to 14 days post last dose in each treatment period
  Number of participants with abnormal vital signs will be assessed.
Number of participants with clinically significant abnormal findings in Electrocardiogram (ECG) Parameters | Up to 14 days post last dose in each treatment period
  Triplicate 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS interval, QT interval, Corrected QT (QTc) interval.
Number of participants with abnormal cardiac telemetry findings | Up to 24 hours post dose on Day 1
  Telemetry is the continuous monitoring of a participants heart rate and rhythm from a remote location. Continuous cardiac telemetry will start in a supine position after at least 5 minutes rest.

SECONDARY OUTCOMES:
Area under the plasma drug concentration (AUC) versus time curve (AUC[0-t]) of GSK3494245 following single dose administration under fasting condition | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 minutes [min], 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate AUC (0-t) of GSK3494245 under fasting condition.
AUC (0-t) of GSK3494245 following single dose administration under fed condition | Cohort 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate AUC (0-t) of GSK3494245 under fed condition.
AUC-time curve from time zero to extrapolated to infinity (AUC[0-inf]) of GSK3494245 following single dose administration under fasting condition | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate AUC (0-inf) of GSK3494245 under fasting condition.
AUC (0-inf) of GSK3494245 following single dose administration under fed condition | Cohort 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate AUC(0-inf) of GSK3494245 under fed condition.
Maximum observed plasma drug concentration (Cmax) of GSK3494245 following single dose administration under fasting condition | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate Cmax of GSK3494245 under fasting condition.
Cmax of GSK3494245 following single dose administration under fed condition | Cohort 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate Cmax of GSK3494245 under fed condition.
Time to maximum observed plasma drug concentration (Tmax) of GSK3494245 following single dose administration under fasting condition | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate Tmax of GSK3494245 under fasting condition.
Tmax of GSK3494245 following single dose administration under fed condition | Cohort 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate Tmax of GSK3494245 under fed condition.
Apparent terminal half-life (t1/2) of GSK3494245 following single dose administration under fasting condition | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate t1/2 of GSK3494245.
t1/2 of GSK3494245 following single dose administration under fed condition | Cohort 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate t1/2 of GSK3494245.
Amount of GSK3494245 excreted in urine over 24 hours (Ae0-24h) following single dose administration | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Urine samples will be collected at the indicated time points to evaluate Ae0-24h of GSK3494245.
Fraction of dose excreted in urine over 24 hours (fe%) of GSK3494245 following single dose administration | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Urine samples will be collected at the indicated time points to evaluate fe% of GSK3494245
Renal Clearance (CLr) of GSK3494245 following single dose administration | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Urine samples will be collected at the indicated time points to evaluate CLr of GSK3494245.
Dose-proportionality assessment using AUC(0-inf) following single dose of GSK3494245 | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate AUC(0-inf) of GSK3494245.
Dose-proportionality assessment using Cmax following single dose of GSK3494245 | Cohort 1, 2 and 3: Day 1 (Pre-dose, 10 min, 30 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12 and 24 hour post dose in each treatment period)
  Blood samples will be collected at the indicated time points to evaluate Cmax of GSK3494245.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com